CLINICAL TRIAL: NCT00608348
Title: Sympathetic Nerve Activity During Hypoglycemia and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Steve Davis, Chairman of Medicine, Vanderbilt University
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: IRB#020777-SNA during hypo/ex
Record Dates: First submitted 2008-01-29; First posted 2008-02-06 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus
Keywords: exercise; hypoglycemia; sympathetic nerve activity
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Hyperinsulinemic euglycemic or hypoglycemic clamp with Muscle and skin sympathetic nerve activity recording in arm and/or leg
  Interventions: Procedure: Hyperinsulinemic glucose clamp procedures
- 2 (Experimental): Exercise with insulin or no insulin infused with muscle and skin sympathetic nerve activity measurements
  Interventions: Procedure: moderate exercise

INTERVENTIONS:
Procedure: Hyperinsulinemic glucose clamp procedures — 2 hours of either euglycemic or hypoglycemic glucose clamping
  Arms: 1
Procedure: moderate exercise — 90 minutes of moderate exercise with either hyperinsulinemia or euinsulinemia
  Arms: 2

SUMMARY:
The purpose of this study is to determine if either hypoglycemia or exercise cause differential responses in muscle and skin sympathetic nerve activity.

DETAILED DESCRIPTION:
The body has defensive responses to correct low blood sugar (hypoglycemia). A vital component of this response is release of glucagon and activation of the sympathetic nervous system, which provides the means for raising blood glucose levels towards normal. We can measure circulating hormones indicating the level of these responses, but additionally, sympathetic nervous system responses can be measured directly. We can measure the sympathetic nerve activity that controls blood flow to muscles (MSNA) and blood flow and sweating to skin (SSNA). The purpose of this study is to determine if either hypoglycemia or exercise cause differential responses in muscle and skin sympathetic nerve activity. We would also like to determine what the sympathetic response is to cycling exercise with insulin and normal blood sugar. Therefore, we would like to test the sympathetic responses to insulin with normal blood glucose, hypoglycemia, and during exercise bouts and normal blood glucose, with or without insulin.

ELIGIBILITY:
Inclusion Criteria:

* 36 Healthy male and female subjects (18 males and 18 females) aged 18-40 yr
* All potential volunteers will have routine blood test to screen for hepatic, renal, and hematological abnormalities
* Body mass index ≤30kg · m-2
* Normal bedside autonomic function
* Female volunteers of childbearing potential will undergo HCG pregnancy test at screening and again on the study day.

Exclusion Criteria:

* Pregnant women
* Subjects unable to give voluntary informed consent
* Subjects on anticoagulant drugs or anemic
* Subjects with a recent medical illness
* Subjects with a history of hypertension, heart disease or cerebrovascular disease
* Subjects with known liver or kidney disease
* Subjects with recent weight loss or consuming a low carbohydrate diet

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2002-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States